CLINICAL TRIAL: NCT00258492
Title: The Prevalence and Outcomes of Restless Legs Syndrome Among Veterans - Exercise Intervention
Brief Title: Restless Legs Syndrome Exercise Intervention
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northeastern Ohio Universities College of Medicine (Other)
Collaborators: Louis Stokes VA Medical Center (U.S. Federal Agency); The University of Akron (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency); Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAMD17-03-1-0082; DAMD17-03-1-0082
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2006-07

CONDITIONS: Restless Legs Syndrome; Insomnia
Keywords: Restless legs syndrome; Insomnia; Daytime sleepiness; Exercise
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence; Motor Activity | interventions — Exercise

INTERVENTIONS:
Behavioral: Aerobic exercise

SUMMARY:
A pilot study of an aerobic exercise intervention to moderate symptoms and improve sleep quality among patients with Restless Legs Syndrome (RLS). We, the researchers at Northeastern Ohio Universities College of Medicine, hypothesize that, relative to a control group, RLS sufferers who participate in an aerobic exercise intervention will demonstrate:

1. reduced RLS symptoms;
2. improved sleep quality;
3. reduced daytime sleepiness.

DETAILED DESCRIPTION:
We will implement an exercise intervention among persons who suffer from RLS.

Study members will be Veterans, over the age of 40, who have been identified as RLS cases as part of our larger study of "The Prevalence and Outcomes of Restless Legs Syndrome among Veterans." We will use a cross-over design in which Veterans will be randomly assigned to the exercise intervention or control. Each arm of the study will be 3 months duration.

The protocol for the intervention will consist of twice weekly supervised exercise sessions. The goal for exercise participants will be to engage in continuous aerobic exercise for 45 minutes at an intensity of approximately 60% of VO2max. The control will be weekly support group meetings.

Outcomes will be measured using standardized sleep scales, actigraphy, and daily sleep and exercise logs.

ELIGIBILITY:
Inclusion Criteria:

* Meets case definition for RLS with symptoms at least one day a week
* Age 40 and older
* Moderate or severe insomnia
* Able to engage in moderate exercise
* Permission of primary care physician to participate in exercise.

Exclusion Criteria:

* Serum ferritin below 50 ng/ml
* Body mass index (BMI) greater than 40
* History of recent myocardial infarction or stroke
* Alcohol use, more than 3 drinks a day
* Current use of medications for sleep

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-12; Study Completion 2007-01

PRIMARY OUTCOMES:
RLS symptom severity, measured bi-weekly

SECONDARY OUTCOMES:
Sleep efficiency, measured bi-weekly
Insomnia severity, measured bi-weekly
Day time sleepiness, measured bi-weekly

CONTACTS AND LOCATIONS:
Overall Officials: Claire C. Bourguet, Ph.D., Principal Investigator — Northeastern Ohio Universities College of Medicine